CLINICAL TRIAL: NCT00054223
Title: Ethics Study To Understand The Decision Making Process Of Phase I Cancer Patients
Brief Title: Study of Decision Making in Patients Participating in Phase I Clinical Trials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None
Other Study IDs: 030063; 03-CC-0063; CDR0000269911
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Psychosocial Effects of Cancer and Its Treatment; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: psychosocial effects of cancer and its treatment; unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Psychiatric Rehabilitation

INTERVENTIONS:
Procedure: psychosocial assessment and care

SUMMARY:
RATIONALE: Studying individuals who are enrolled in phase I clinical trials may help to improve the way in which clinical trials are conducted.

PURPOSE: This clinical trial is studying patients' personality traits, reasons for participating in the trial, and understanding of their medical situation, prognosis, and risks and benefits of participating in a phase I trial.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the range of personality traits of patients enrolled in a phase I clinical trial.
* Determine these patients' understanding of their medical situation and prognosis.
* Determine these patients' understanding of risks and benefits of phase I clinical trials.
* Determine these patients' reasons for participating in a phase I clinical trial.
* Determine the risk/benefit trade-offs of these patients.
* Determine the existential outlook of these patients.
* Determine the information gathering nature of these patients.

OUTLINE: This is a multicenter study.

Before beginning phase I clinical trial treatment, patients complete a survey over 30-45 minutes administered by an interviewer. Patients then self-administer the Temperament and Character Inventory assessment over 30 minutes.

PROJECTED ACCRUAL: Approximately 250 patients will be accrued for this study within 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Consented to enrollment in a phase I cancer clinical trial

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Understands written English

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No concurrent enrollment in other clinical trials evaluating phase I patient attitudes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2003-01; Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manish Agrawal, MD, Study Chair — National Cancer Institute (NCI)
Locations (5):
- United States (5):
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Cancer Therapy and Research Center, San Antonio, Texas